CLINICAL TRIAL: NCT01408511
Title: A Multicenter, Open Label Study to Evaluate the Adrenal Suppression Potential of Mapracorat 0.1% Ointment in Adults With Atopic Dermatitis
Brief Title: HPA Axis Study in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15446; 1403161 (Other: Company Internal)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Mapracorat

INTERVENTIONS:
Drug: Mapracorat — Application of the investigational product on the affected skin areas

SUMMARY:
A multicenter, open-label study to evaluate the adrenal suppression potential of Mapracorat 0.1% ointment in adults with atopic dermatitis.

DETAILED DESCRIPTION:
Assessment of safety, efficacy, pharmacokinetics and adrenal suppression potential of Mapracorat 0.1% ointment in adults with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female subject aged >= 18 years
* Diagnosis of atopic dermatitis according to Hanifin and Rajka Criteria
* Investigator's Global Assessment (IGA) score of 3 (moderate) to 4 (severe) at baseline
* Normal ACTH response before start of treatment

Exclusion Criteria:

* Pregnancy or lactation
* Clinically relevant disease, which could interfere with the study conduct or the evaluation and interpretation of the study results
* Concomitant medical or dermatological disorder(s), which could interfere with the study conduct or the evaluation and interpretation of the study results
* Clinically manifest immunosuppressive disorder or known history of malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-21 (Actual)

PRIMARY OUTCOMES:
HPA axis response to Cosyntropin: Number of subjects with adrenal suppression | measured after 4 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- South Africa (3):
  - PAREXEL Bloemfontein, Bloemfontein
  - PAREXEL George, George
  - PAREXEL Port Elizabeth, Port Elizabeth